A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study to Compare Perrigo UK FINCO Clindamycin Phosphate and Benzoyl Peroxide Topical Gel 1.2%/3.75% to Valeant Pharmaceuticals North America, LLC Onexton™ Topical Gel (Clindamycin Phosphate and Benzoyl Peroxide Gel 1.2%/3.75%), and Both Active Treatments to a Vehicle Control in the Treatment of Acne Vulgaris

NCT02515305

06-12-2015

# STATISTICAL ANALYSIS PLAN

Clindamycin Phosphate and Benzoyl Peroxide Topical Gel 1.2%/3.75% Protocol PRG-NY-15-003



A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study to Compare Perrigo UK FINCO Clindamycin Phosphate and Benzoyl Peroxide Topical Gel 1.2%/3.75% to Valeant Pharmaceuticals North America, LLC Onexton™ Topical Gel (Clindamycin Phosphate and Benzoyl Peroxide Gel 1.2%/3.75%), and Both Active Treatments to a Vehicle Control in the Treatment of Acne Vulgaris



# **Table of Contents**

| 1 | Purpose of Statistical Analysis Plan | | |
|---|---|---|---|
| 2 | Stu | Study Objectives | |
| 3 | Stu | dy Design | 4 |
| 4 | Pop | oulations To Be Analyzed | 5 |
| 5 | Pla | nned Analyses | 6 |
| | 5.1 | Methodological Considerations | |
| | 5.2 | | |
| | | Handling of Dropouts or Missing Data | |
| | 5.3 | Demographics and Baseline Characteristics | 6 |
| | 5.4 | Subject Accountability | 7 |
| | 5.5 | Efficacy Variables and Analyses | 7 |
| | 5.5. | J T | |
| | 5.5. | · 1 | |
| | 5.5. | | |
| | 5.6 | Safety Variables and Analyses | 9 |
| 6 | App | Appendices | |
| | 6.1 | Handling of Missing or Incomplete Dates for Adverse Events and Concomitant Medications | 10 |
| | 6.2 | Summary of Assessments | 10 |
| 7 | Tab | oles and Listings | . 12 |
| | | ble 14.1.1- Subject Final Study Disposition | |
| | | ble 14.1.2- Subject Enrollment and Protocol Violations | |
| | | ble 14.1.3- Subject Enrollment by Study Site | |
| | | ble 14.1.4.1- Demographic Characteristics for Intent-to-Treat Population | |
| | | ble 14.1.4.2- Demographic Characteristics for Modified Intent-to-Treat Population | |
| | | ble 14.1.4.3- Demographic Characteristics for Per-Protocol Population | |
| | | ole 14.1.5.2- Baseline Vital Signs for Modified Intent-to-Treat Population | |
| | | ble 14.1.5.3- Baseline Vital Signs for Per-Protocol Population | |
| | | ole 14.2.1.1- Primary Efficacy Analysis: Mean Percent Change Baseline <sup>3</sup> to Week 12 (Visit 4/Day 84) in | |
| | | Number of Inflammatory Lesion Counts | |
| | | ole 14.2.1.2- Primary Efficacy Analysis: Mean Percent Change from Baseline <sup>3</sup> to Week 12 (Visit 4/Day 84) Jumber of Non-Inflammatory Lesion Counts | |
| | | ble 14.2.2- Secondary Efficacy Analysis: Proportion of Subjects with Clinical Success on the Investigator's | . 22 |
| | G | Global Assessment (IGA) at Week 12 (Visit 4/Day 84) | 23 |
| | | ble 14.2.3.1- Additional Efficacy Summary: Post-Baseline Inflammatory Lesion Count for Per-Protocol | 2.4 |
| | | opulationble 14.2.3.2- Additional Efficacy Summary: Post-Baseline Inflammatory Lesion Count for Modified Intent-t | |
| | | reat Population | |
| | Tab | ole 14.2.3.3- Additional Efficacy Summary: Post-Baseline Non-Inflammatory Lesion Count for Per-Protoco | l |
| | | Population | . 25 |
| | | ble 14.2.3.4- Additional Efficacy Summary: Post-Baseline Non-Inflammatory Lesion Count for Modified Intent-to-Treat Population | 25 |
| | Tab | ole 14.2.3.5- Additional Efficacy Summary: Post-Baseline Investigator's Global Assessment (IGA) and | |
| | C | Clinical Success for Per-Protocol Population | 26 |

| Table 14.2.3.6- Additional Efficacy Summary: Post-Baseline Investigator's Global Assessment (IG Clinical Success for Modified Intent-to-Treat Population | |
|---|---|
| Table 14.3.1- Duration of Treatment and Medication Compliance Rate for Intent-to-Treat Population | |
| Table 14.3.2.1- Overall Summary of Treatment Emergent Adverse Events (TEAEs) for Intent-to-Treatment Emergent Adverse Events (TEAEs) for Intent-to-Treatment Emergent Adverse Events (TEAEs) for Intent-to-Treatment Emergent Adverse Events (TEAEs) for Intent-to-Treatment Emergent Emergent Events (TEAEs) for Intent-to-Treatment Events (TEAEs) for Intent-to-Treatment E | reat Popula |
| Table 14.3.2.2- Summary of Treatment-Emergent Adverse Events (TEAEs) by MedDRA System C | Organ Clas |
| Preferred Term for Intent-to-Treat Population | |
| Table 14.3.2.3- Summary of Treatment-Emergent Adverse Events (TEAEs) by MedDRA System C | Organ Clas |
| Preferred Term, and Severity for Intent-to-Treat Population | |
| Table 14.3.2.4- Summary of Treatment-Emergent Adverse Events (TEAEs) by MedDRA System C<br>Preferred Term, and Relationship to Study Medication for Intent-to-Treat Population | |
| Table 14.3.2.5- Summary of Skin Related Treatment-Emergent Adverse Events (TEAEs) by MedD Organ Class and Preferred Term for Intent-to-Treat Population | |
| Table 14.3.2.6- Common Treatment-Emergent Adverse Events (TEAEs) by MedDRA System Organ Preferred Term for Intent-to-Treat Population | |
| Table 14.3.3.1- Application Site Reaction Assessment (Erythema) by Visit for Intent-to-Treat Popu | |
| Table 14.3.3.2- Application Site Reaction Assessment (Dryness) by Visit for Intent-to-Treat Popular | |
| Table 14.3.3.3- Application Site Reaction Assessment (Scaling/Peeling) by Visit for Intent-to-Treat | |
| Table 14.3.3.4- Application Site Reaction Assessment (Burning/Stinging) by Visit for Intent-to-Tre | |
| Table 14.3.3.5- Application Site Reaction Assessment (Erosion) by Visit for Intent-to-Treat Popula | |
| Table 14.3.3.6- Application Site Reaction Assessment (Edema) by Visit for Intent-to-Treat Populat | ion |
| Table 14.3.3.7- Application Site Reaction Assessment (Pain) by Visit for Intent-to-Treat Population | 1 |
| Table 14.3.3.8- Application Site Reaction Assessment (Itching) by Visit for Intent-to-Treat Populat | ion |
| ct Listings | |
| Listing 16.2.1.1- Subject Analysis Status | |
| Listing 16.2.1.2- Subject End-of-Study Status | |
| Listing 16.2.1.3- Date of Visit | |
| Listing 16.2.2.1- Protocol Violations and Deviations | |
| Listing 16.2.2.2- Comments | |
| Listing 16.2.2.3- Inclusion/Exclusion Criteria | |
| Listing 16.2.4.1- Demographics and Informed Consent at Baseline | |
| Listing 16.2.4.2- Vital Signs at Baseline | |
| Listing 16.2.4.3- Brief Physical Examination (With Abnormality Only) | |
| Listing 16.2.4.4- Subject Medical History (With Past or Current Findings) | |
| Listing 16.2.5.1- Study Medication/ Diary Card Dispensing | |
| Listing 16.2.5.2- Subject Compliance During Study | |
| Listing 16.2.5.3- Telephone Contact | |
| Listing 16.2.5.4- Treatment Record | |
| Listing 16.2.5.5- Subject Compliance at End of Study | |
| Listing 16.2.6.1- Dermatological Assessment and Investigator's Global Assessment (IGA) | |
| Listing 16.2.6.2- Efficacy Response for Per-Protocol Population | |
| Listing 16.2.6.3- Efficacy Response for Modified Intent-to-Treat Population | |
| Listing 16.2.7.1- Adverse Events | |
| Listing 16.2.7.2- Adverse Events Leading to Study Treatment Interruption/Discontinuation | |
| Listing 16.2.7.3- Serious Adverse Events | |
| Listing 16.2.8.1- Urine Pregnancy Test (Female Subjects Only) | |
| Listing 16 2.0.1 Application City Departure Assessment | |
| Listing 16.2.9.1- Application Site Reaction Assessment | |

Perrigo, Inc.
SAP Version: 1.0
Protocol: PRG-NY-15-003

# **List of Abbreviations**

| AE | Adverse Event |
|----------|----------------------------------------------|
| ANOVA | Analysis of Variance |
| CI | Confidence Interval |
| CMH | Cochran-Mantel Haenszel Test |
| IGA | Investigator's Global Assessment |
| ITT | Intent-to-Treat (Population) |
| LOCF | Last Observation Carried Forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | Modified Intent-to-Treat (Population) |
| PD | Protocol Deviation |
| PP | Per-Protocol (Population) |
| PV | Protocol Violation |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| TEAE | Treatment-Emergent Adverse Event |
| TESAE | Treatment-Emergent Serious Adverse Event |
| WHO Drug | World Health Organization Drug Dictionary |

Perrigo, Inc.
Protocol: PRG-NY-15-003
SAP Version: 1.0

### Statistical Analysis Plan

# 1 Purpose of Statistical Analysis Plan

The purpose of the statistical analysis plan is to describe in detail all the data, statistical methods, and summary tables required to implement the statistical analysis of Clinical Study Protocol PRG-NY-15-003

## 2 Study Objectives

To compare the safety and efficacy profiles of Perrigo UK FINCO Clindamycin Phosphate and Benzoyl Peroxide Topical Gel 1.2%/3.75% to Valeant Pharmaceuticals Onexton™ Topical Gel (Clindamycin Phosphate and Benzoyl Peroxide Gel 1.2%/3.75%) and to demonstrate the superior efficacy of the two active formulations over that of the vehicle in the treatment of acne vulgaris.

## 3 Study Design

For the purpose of exploring the above objectives, the study will be conducted as a double-blind, randomized, parallel-group, vehicle-controlled, multicenter trial.

| Approximately healthy males and females, 12 to 40 years of age, inclusive, who meet the |
|---|
| inclusion/exclusion criteria, will be enrolled to obtain approximately modified-Intent-To |
| Treat (mITT) and per-protocol (PP) subjects. |

The actual number of subjects enrolled in the study will be based on blinded review of subject status (related to the per-protocol definition, section 4) to determine that the number of subjects expected to meet the PP criteria is sufficient.

If this number is expected to be met prior to enrolling subjects, the enrollment will be closed.

Each subject will be randomly assigned to one of following treatment groups in a

(1) Test: Clindamycin Phosphate and Benzoyl Peroxide Topical Gel 1.2%/3.75%,

(2) Reference: Onexton™ Topical Gel (Clindamycin Phosphate and Benzoyl Peroxide Gel 1.2%/3.75%), Valeant Pharmaceuticals North America, LLC

(3) Vehicle of test product Perrigo UK FINCO,

Subjects will be admitted into the study only after written informed consent has been obtained and all of the inclusion and none of the exclusion criteria have been met. Randomization will be performed according to a computer generated randomization scheme where the treatment group designation has been assigned to the subject number. The treatment designation will remain blinded until the final database is closed. An independent third party generator will generate and hold the randomization code throughout the study. Randomized subjects will apply study medication onto six areas of the face (chin, left cheek, right cheek, nose, left forehead and right forehead) avoiding contact with the eyes, lips, mouth, broken areas of the skin and mucous membranes at approximately the same time once daily for 12 weeks.

Subjects will be scheduled for an office visit for Visit 1/Day 1 (Baseline), Visit 2/Week 4/Day 28 (±4 days)(Interim, Visit 3/Week 8/Day 56 (±4 days)(Interim), and Visit 4/Week 12/Day 84 (±4 days) (End of treatment/End of study). Safety will be assessed by monitoring adverse events at each visit and at the Week 2/Day 15 (±4 days) Telephone Contact.

## 4 Populations To Be Analyzed

Three subject populations are defined as follows:

- (1) <u>Intent-to-Treat (ITT) (safety population)</u>: Any subject that was randomized, received and used study medication;
- (2) <u>Modified Intent-to-Treat (mITT)</u>: Any subject, who met the inclusion/exclusion criteria, was randomized, received and used the study medication, and returned for at least one post-baseline efficacy assessment;
- (3) Per-Protocol (PP): Any subject:
  - Who met inclusion/exclusion criteria,
  - Who was randomized and received and used study medication,
  - Who met the protocol criteria for compliance
     and
  - Who completed Visit 4/Week 12/Day 84 (End of Treatment/Early Termination Visit) within window OR was dropped from the study due to treatment failure treatment
  - Without significant protocol violations that could have interfered with the administration of the treatment or the precise evaluation of treatment efficacy.





### 5 Planned Analyses

#### 5.1 Methodological Considerations

The study will be conducted under the same protocol across all the sites. No formal statistical analyses are planned to evaluate the consistency of efficacy results across the multiple clinical sites. These results, however, will be tabulated and if a site's efficacy data are obviously inconsistent with the results across all sites, this will be explored and addressed in the final study report.

Two-sided hypothesis testing will be conducted for all the tests. Resulting p-values less than 0.05 will be considered statistically significant unless noted otherwise. No adjustments of p-values for multiple comparisons will be made. No interim analyses are planned. SAS software will be used for all data analyses and tabulations.



#### 5.3 Demographics and Baseline Characteristics

Baseline variables (e.g., sex, age, ethnic origin) will be evaluated, adjusting for site, to identify differences between treatment groups, which were not eliminated by randomization. Any significant baseline differences will be reviewed for their potential impact on the efficacy findings.

Continuous variables at baseline will be examined by two-way analysis of variance (ANOVA) with treatment and site as fixed effects when normal error and homogeneous variance assumptions are satisfied, or by the nonparametric rank based ANOVA when they are not, to compare treatment group differences.

Categorical variables such as gender, race, etc., will be examined by Cochran-Mantel-Haenszel test, stratified by site.

Summary tables by treatment group will be presented. For each continuous variable, the summary will include the mean, standard deviation, minimum and maximum. For each categorical variable, the summary will include frequencies and percentages.

# 5.4 Subject Accountability

A summary of subject disposition will be provided for all subjects. Descriptive summaries of subject disposition, reason for discontinuation, and analyses population will be provided by treatment group. The data will also be presented in subject data listings.

## 5.5 Efficacy Variables and Analyses

# 5.5.1 Primary Endpoints

The primary efficacy endpoints are the mean percent change from baseline to Week 12 (Visit 4/Day 84) in the inflammatory (papules and pustules) lesion counts AND the mean percent change from baseline to Week 12 (Visit 4/Day 84) in the non-inflammatory (open and closed) lesion counts.

#### Equivalent Efficacy

For the mean percent change from baseline in the inflammatory lesion counts, the Test treatment will be considered to be therapeutically equivalent to the Reference treatment if the 90% confidence interval on the Test-to-Reference ratio of means, calculated by Fieller's Method, falls within the interval 0.80 to 1.25. The compound hypothesis to be tested for therapeutic equivalence between test and reference is:

$$H_0: \mu_T/\mu_R \le 0.80 \text{ or } \mu_T/\mu_R \ge 1.25 \text{ versus}$$

$$H_{_{\mbox{\scriptsize A}}}\!\!: 0.80 < \mu_{_{\mbox{\scriptsize T}}}/\mu_{_{\mbox{\scriptsize R}}} < 1.25.$$

Where  $\mu_T$  and  $\mu_R$  are the mean percent change from baseline to Week 12 (Visit 4/Day 84) in inflammatory lesions counts for the test treatment and the reference treatments, respectively. The null hypothesis is rejected when the two-sided 90% confidence interval (CI) for the ratio of means between test and reference products is between 0.80 and 1.25. Rejection of the null hypothesis supports the conclusion of therapeutic equivalence between test and reference products for the primary efficacy variable.

The two-sided 90% confidence interval will be constructed using an ANOVA model adjusting for the effects of treatment and site.

The same analysis will be applied to the mean percent change from baseline in the non-inflammatory lesion count.

Therapeutic equivalence evaluations in the per-protocol (PP) population will be considered definitive and those in the mITT will be considered supportive.

### Superiority

For the percent change from baseline in the inflammatory lesion counts, each active treatment will be evaluated to determine if it has superior efficacy to that of the Vehicle at Week 12 (Visit 4/Day 84) via ANOVA model containing terms for treatment and site. The compound hypothesis to be tested for superiority of test and reference over Vehicle is:

$$\boldsymbol{H}_{\!0}\!:\boldsymbol{\mu}_{\!T}\!\leq\!\boldsymbol{\mu}_{\!V}\,\text{or}\;\boldsymbol{\mu}_{\!R}\!\leq\!\boldsymbol{\mu}_{\!V}\,\text{versus}$$

$$H_A$$
:  $\mu_T > \mu_V$  and  $\mu_R > \mu_V$ 

Where  $\mu_T$ ,  $\mu_R$  and  $\mu_V$  are the mean percent change from baseline to Week 12 (Visit 4/Day 84) in inflammatory lesions counts for the test, the reference and the vehicle treatments, respectively. The null hypothesis is rejected when both p-values from the ANOVA are less than 0.05 (two-sided test). Rejection of the null hypothesis supports the conclusion of superiority of test and reference products over the vehicle product for the primary efficacy variable.



#### 5.5.2 Secondary Endpoint

The secondary efficacy endpoint is the proportion of subjects with clinical success on the Investigator's Global Assessment (IGA) at Week 12 (Visit 4/Day 84), where success is defined as an IGA score that is at least 2 grades less than the baseline assessment.

#### Equivalent Efficacy

The Test treatment will be considered to be therapeutically equivalent to the Reference treatment if the 90% Wald confidence interval with Yates' continuity correction on the difference in their success proportions is contained within the interval of -20% to +20%.

#### Superiority

The proportion of subjects with clinical success for each active treatment will be compared separately between each of the active treatments and the Vehicle using two-sided,  $\alpha = 0.05$ , continuity-corrected Z-tests.

Equivalence and superiority analyses will be conducted in both the PP and mITT populations.



### 5.6 Safety Variables and Analyses

#### Duration of Treatment and Medication Compliance

Number of applications, days of exposure, and compliance rate will be summarized by treatment group using descriptive statistics. For each subject, the overall duration of treatment (days) will be calculated using the following formula:

(Date of last application of study medication) - (Date of first application of study medication) + 1.

Medication compliance rate (%) will be calculated for each subject as follows:

(Total number of applications used) / (Expected number of applications) \*100%.



## Adverse Events

Adverse events (AEs) will be coded in MedDRA, version 15.1. Treatment-Emergent Adverse Event (TEAE) is defined as any AE occurs on or after applying the first dose of study drug. Number and percent of subjects reporting TEAEs will be tabulated by treatment group. Summaries will be presented by body system and preferred term for the ITT population. Similar tables will be presented by severity and relationship to study drug. TEAEs reported by more than 5% subjects for any treatment group will also be summarized. In summaries of incidence rates (frequencies and percentages), severity and relationship to study drug, subjects who report more than one event that are mapped to the same preferred term will be counted only once under the strongest severity and relationship, accordingly. The difference between Test and Reference treatments with regard to the severity and frequency of their dermatological adverse events wil be statistically evaluated. Fisher's exact test will be used to compare the proportions of subjects of the two active treatment groups who report any TEAE.

Treatment-Emergent Serious Adverse Events (TESAEs) and TEAEs that led to treatment interruption or discontinuation will be presented in data listings.

## **Concomitant Medications**

Concomitant medications will be coded using the WHO Drug Dictionary, version September, 2014, and will be presented in data listings.

#### **Application Site Reactions**

Perrigo, Inc.
Protocol: PRG-NY-15-003
SAP Version: 1.0

Frequency and distribution of application site reactions of erythema, dryness, scaling/peeling, burning/stinging, erosion, edema, pain and itching will be summarized and compared descriptively by visit.

Safety comparisons will be performed only for the ITT population.

# 6 Appendices

6.1 Handling of Missing or Incomplete Dates for Adverse Events and Concomitant Medications

#### Adverse Events

Handling of partial dates is only considered for the start date. An adverse event with a partial start date is considered treatment emergent if:

- only the day is missing and the start month/year is the same or after the month/year of the first dose
- the day and month are missing and the start year is the same or greater than the year of the first dose date
- the start date is completely missing

## **Concomitant Medications**

Handling of partial dates is only considered for the stop date. A medication with a partial stop date is considered concomitant if:

- only the day is missing and the stop month/year is the same or after the month/year of the first dose
- the day and month are missing and the stop year is the same or greater than the year of the first dose date
- the stop date is completely missing or the medication is ongoing

## 6.2 Summary of Assessments

The schedule of visits and procedures to be conducted at each visit are summarized in the Schedule of Study Procedures.

Perrigo, Inc. SAP Version: 1.0 Protocol: PRG-NY-15-003

